CLINICAL TRIAL: NCT02407886
Title: Retinal Ganglion Cell Layer in Patients With Intracerebral Processes
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-0649
Record Dates: First submitted 2015-03-05; First posted 2015-04-03 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Ganglion Cells

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Transsynaptic degeneration of the retinogeniculate pathways is well documented to occur in nonhuman primates when the cerebral lesion occurs even during adulthood. In case of humans, retrograde transsynaptic degeneration of the retinogeniculate pathways has been shown to occur following prenatal or perinatal lesions, but its occurrence after cerebral lesions in adults is considerable rare. It is, however, well established that retrograde transsynaptic degeneration affects other neural systems in humans even when the injury occurs during adulthood. Some histopathological evidence points to the possibility of transsynaptic degeneration of the retinogeniculate pathway in humans even when the lesion occurs in adults, but the clinical significance is unknown.'

Purpose:

To measure the retinal ganglion cell layer (GCL) in patients with visual field defects due to intracerebral processes. To correlate GCL with the localization and type of intracerebral lesion.

To compare the GCL with the retinal nerve fibre layer (RNFL) to investigate, which of the 2 parameters is more sensitive to show retinal layer abnormalities.

To correlate GCL with visual field defects and electrophysiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with intracerebral lesions within the central visual tract
* associated visual field defects
* investigations (OCT, ERG) possible

Exclusion Criteria:

* lesions within the optic nerve without extension in the optic tract
* neurological disease
* optic disc anomalies: glaucoma, nystagmus, high myopia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with intracerebral lesions
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Ganglion cell thickness | measurements will be taken at a minimum of 4 weeks after the inital diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Christina Gerth-Kahlert, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland